CLINICAL TRIAL: NCT02145949
Title: Mechanistic Approach to Preventing Atrophy and Restoring Function in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Slocum Center for Orthopedics and Sports Medicine (Other); Slocum Research & Education Foundation (Other); Oregon Research Institute (Other); Oregon Health and Science University (Other); University of Arkansas (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hans Dreyer, Assistant Professor, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12272013.024; R01AG046401 (NIH)
Record Dates: First submitted 2014-05-19; First posted 2014-05-23 (Estimated); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Muscle Atrophy; Quality of Life
Keywords: aging; clinical; translational; functional mobility; total knee arthroplasty
MeSH Terms: conditions — Muscular Atrophy | interventions — Amino Acids, Essential; Histidine; Isoleucine; Leucine; Methionine; Phenylalanine; Threonine; Valine; Tryptophan; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Essential Amino Acids (EAA) (Experimental): Aim 1: Twice-daily ingestion of 20 g of EAA for 1 wk before through 6 wk after TKA.
  Supplement composition for the EAAs: histidine, 2.2 g (11% of total); isoleucine, 2.0 g (10%); leucine, 3.6 g (18%); lysine, 3.2 g (16%); methionine, 0.6 g (3%); phenylalanine, 3.2 g (16%); threonine, 2.8 g (14%); and valine, 2.4 g (12%).
  Aim 2: Twice-daily ingestion of 23 g of EAA for 1 wk before through 6 wk after TKA.
  Supplement composition for the EAAs: histidine, 1.28 g (5% of total); isoleucine, 1.8 g (8%); leucine, 7.4 g (32%); lysine, 3.6 g (15%); methionine, 1.76 g (8%); phenylalanine, 3.1 g (13%); threonine, 1.9 g (8%); valine, 2.08 g (9%); and tryptophan, 0.5 g (2%).
  Interventions: Drug: Essential Amino Acids (EAA)
- Placebo (Alanine) (Placebo Comparator): Aim 1: Twice-daily ingestion of 20 g of Alanine (Non-essential amino acid) for 1 wk before through 6 wk after TKA.
  The placebo supplement consists of 20 g (100%) alanine.
  Aim 2: Twice-daily ingestion of 23 g of Alanine (Non-essential amino acid) for 1 wk before through 6 wk after TKA.
  The placebo supplement consists of 23 g (100%) alanine.
  Interventions: Drug: Placebo (Alanine)

INTERVENTIONS:
Drug: Essential Amino Acids (EAA) — Twice daily ingestion of 20 or 23 grams of EAA for 7 days leading up to surgery and continuing for 6 weeks after surgery [surgery = primary total knee arthroplasty]
  Other Names: L-Histidine; L-Isoleucine; L-Leucine; L-Lysine monohydrochloride; L-Methionine; L-Phenylalanine; L-Threonine; L-Valine; L-Tryptophan
  Arms: Essential Amino Acids (EAA)
Drug: Placebo (Alanine) — Twice daily ingestion of 20 or 23 grams Placebo (alanine) for 7 days leading up to surgery and continuing for 6 weeks after surgery [surgery = primary total knee arthroplasty]
  Other Names: L-Alanine, A4349 (Non-essential amino acid)
  Arms: Placebo (Alanine)

SUMMARY:
As a function of the growing population of older adults, an estimated 3.48 million total knee arthroplasty (TKA) procedures will be performed annually in the U.S. by 2030. Despite the near-universal success of this surgery in mitigating chronic knee pain, TKA is not successful in restoring long-term physical function in older adults, primarily because of quadriceps muscle atrophy, which explains 77% of the strength deficits. Overall, strength and functional mobility in TKA patients is 30-50% below age-matched healthy controls. Functional tasks such as stair-climbing remain a clinical problem for 75% of patients following TKA. Muscle atrophy occurs in both operative and non-operative legs, and is essentially permanent for older patients because of their impaired ability to increase muscle mass. The purpose of this clinical research is to determine the effects of essential amino acid (EAA) supplementation on muscle mass, strength, and functional mobility following TKA in older adults. Based on strong preliminary data, the investigators hypothesize that twice-daily ingestion of 23 g of EAA for 1 wk before through 6 wk after TKA will increase basal rates of muscle protein synthesis via inactivation of catabolic signaling, and up-regulation of anabolic and cyto-protective proteins. The investigators further hypothesize that short-term atrophy prevention and accelerated return of functional mobility will lead to longer-term structural and functional adaptations, and improved quality of life in older TKA patients vs. Placebo. Identifying the mechanisms up-regulated by EAA treatment that preserve muscle volume and mobility will have a major impact on rehabilitation science. This study will accomplish two specific aims: (1) determine if EAA elevates basal rates of muscle protein synthesis by up-regulating anabolic pathways and cyto-protective proteins, and inactivating catabolic pathways in the short term vs. Placebo and (2) determine if short-term prevention of atrophy, weakness, and functional mobility leads to positive changes in muscle cell structure and function, and improved quality of life in the longer term vs. Placebo. This work is significant because it advances knowledge of the molecular and cellular changes occurring during muscle atrophy (Placebo) and atrophy prevention (EAA) in a clinical setting using a treatment that is broadly applicable, is well tolerated, and can be implemented immediately.

DETAILED DESCRIPTION:
The investigative team has completed recent studies showing that essential amino acid (EAA) supplementation attenuates quadriceps atrophy and accelerates the return of functional mobility following TKA. For patients on EAA, quadriceps atrophy was only -6% and -3% in the operative and non-operative quadriceps, respectively, 6 wks after TKA, but -18% and -10%, respectively, in patients on Placebo, a threefold difference. Of clinical relevance, the patients on EAA were able to maintain strength and demonstrated an accelerated return of functional mobility vs. Placebo 6 wks post-TKA. Positive changes at the cellular level are likely responsible for the reduction in muscle loss and preservation of strength, and to explain the acceleration of the return of functional mobility. As such, we hypothesize that twice-daily ingestion of 23 g of EAA from 1 wk before to 6 wks after TKA will increase basal rates of muscle protein synthesis via inactivation of catabolic signaling (FoxO3a), and up-regulation of anabolic and cyto-protective proteins. We also propose that short-term atrophy prevention and accelerated return of functional mobility will translate into long-term (6 mo and 1 yr post-TKA) structural and functional adaptations, leading to improved quality of life in TKA patients with EAA supplementation vs. Placebo.

The study will use a two-arm parallel design to determine the effect of EAA supplementation on post-TKA muscle cell structure and function, and quality of life in the shorter term (6 months post-TKA) and long term (1 yr post-TKA) vs. Placebo. Subjects will be 80 older male and female adults having primary TKA at the Slocum Center for Orthopedics and Sports Medicine, Eugene, Oregon. Slocum study staff will pre-screen/identify potential subjects for recruitment based on inclusion/exclusion criteria. Eligible patients will be invited to join the study. After the completion of informed consent procedures, participants will be assigned a unique patient identification number, and randomly assigned to either EAA or Placebo on a 1:1 allocation ratio, with blinding of treatment condition to subject and research staff/statisticians collecting data. Twice-daily ingestion of 23 g of supplement will begin 7 days prior to TKA and end at 6 wks post. EAA subjects will receive EAA and Placebo subjects will receive the non-essential amino acid Alinine. Subjects will document compliance with the supplement protocol in a log book and will return empty vials. Subjects will be followed for 1 yr.

Key research questions are: (a) Does EAA prevent shorter-term (6 wks post-TKA) bilateral muscle atrophy, preserve quadriceps strength, and accelerate the return of functional mobility vs. Placebo? (b) Are there shorter-term sex differences on outcome measures? (c) Will EAA increase longer-term (6 mo post-TKA) quadriceps strength and functional mobility vs. Placebo? (d) Does EAA improve long-term (1 yr post-TKA) functional mobility and measures of quality of life vs. Placebo? (e) Are there long-term sex differences in functional mobility or measures of quality of life? Assessment points will be at 6 wks, 4 wks, and 1 wk prior to surgery, and 1 wk, 2 wks, 6 wks, 6 mos, and 1 yr post-TKA. At different assessment points, we will collect demographic, medical (e.g., length of hospital stay, tourniquet use), physiological (e.g., muscle biopsy, MRI, DEXA, strength; blood tests), pharmacologic, functional mobility, physical activity (accelerometer), psychometric (e.g., quality of life; Veterans RAND 12-item Health Survey [VR-12]), food intake (3-day diary), physical therapy, and perceived pain data. The following schedule of assessments will be followed: no more than 6 mo pre-TKA (enrollment and screening), 6 wks pre-TKA (screening, surveys, DEXA scan, MRI test, physical activity and food recording), 4 weeks pre-TKA (blood draw, strength and functional mobility testing, muscle and fat biopsy); 1 wk pre-TKA and in hospital (physical activity and food recording); 1 wk post-TKA (physical activity and food recording); 2 wks post-TKA (blood draw, physical activity and food recording); 6 wks post-TKA (blood draw, MRI test, strength and functional mobility testing, physical activity and food recording, muscle and fat biopsy); 3 mos post-TKA (surveys, strength and functional mobility testing, physical activity and food recording); 6 mos post-TKA (surveys, DEXA scan, MRI test, strength and functional mobility testing, physical activity and food recording, muscle and fat biopsy), and 1 yr (surveys, DEXA scan, MRI test, strength and functional mobility testing, physical activity and food recording, muscle and fat biopsy).

Data will be collected from a variety of sources, including surveys, electronic medical records, medical and functional tests, and staff reports. Data will be entered and double-verified in password-protected spreadsheets sand databases stored behind a firewall. Any electronic medical records data captured will use secure data transfer and HIPAA-compliant protocols approved by the University of Oregon IRB. Staff reports will be forwarded directly to project data managers. All personal data will be identified by numbers rather than names. Interim reports of project results will be made to the Data and Safety Monitoring Board.

Power analyses indicated that a sample size of 80 subjects would be sufficient to detect anticipated effects on primary outcomes: operative leg quadriceps volume (MRI), non-operative leg quadriceps volume (MRI), isometric strength, Get Up And Go test, stair climb up test, stair climb down test, and six-minute walk test. The mean effect size across these outcomes, based on baseline- to 6-week percent change in pilot data) was d = 1.01, reflecting large effects. For a sample size of 30/group, this study can detect ESs of d > .79 with 85% power, and the minimally detectable ES drops to 0.68 or 0.52 with pretest covariates of r = .50 or .75. Every effort will be made to reduce attrition and obtain data on all participants at all assessment points. However, attrition is expected. Because this study will have power to detect anticipated physiological and functional effects with 30 subjects per condition, we will enroll 80 total subjects (40/condition) to account for possible attrition.

The EAA intervention is designed to attenuate muscle loss, improve functional outcomes, and enhance quality of life. Data analyses will focus on shorter-term, longer-term results, and change over time. Preliminary analyses will employ descriptive statistics to understand the nature of the data and ensure that data distributions are appropriate for the statistical tests employed. Chi-square tests and analyses of variance, as appropriate, will be conducted to evaluate the equivalence of continuing participants vs. dropouts on demographic, medical history, and recent levels of dependent variables.

We will conduct random coefficients analysis (RCA) to model muscle and functional mobility across time, as well as covariates that could affect outcomes, such as age, sex, physical activity, and dietary intake. RCA models trajectories from assessments nested within subjects; test of condition are represented by the interaction between a time factor and treatment condition. The RCA avoids the many pitfalls associated with traditional repeated measures ANOVA: It adjusts for within-individual dependence or autocorrelation in the data, can model nonlinear growth, does not require fixed spacing among assessments, and accommodates missing values over time. By using any available data across time, the RCA will limit the effects of missing data, reducing bias and increasing power. Based on our preliminary data, we estimate that we will be able to collect >92% of all data points.

Expected study outcomes are as follows:

1. With successful completion of this research, we expect to demonstrate that EAA prevents muscle atrophy bilaterally, as our preliminary data suggest. To date, it is not known if EAA can prevent atrophy.
2. We expect to show that atrophy prevention will lead to strength gains and accelerated return of functional mobility. We further expect to show that EAA may have positive effects on central activation deficits, as our preliminary data suggest that strength is increased by 6 wks with EAA. To date, it is not known if preserving muscle following TKA will increase strength and augment the return of functional mobility.
3. We expect to document that EAA will increase muscle cell size (CSA) bilaterally, in the vastus lateralis of the operative and non-operative quadriceps. It is not known if atrophy prevention and early return of functional mobility will stimulate positive gains in muscle cell structure.
4. We expect to demonstrate that EAA increases mitochondrial mass bilaterally and increases mitochondrial respiration at rest. By sampling from the non-operative (control leg) and operative leg, we expect to show that EAA normalizes mitochondrial function over time (6 mo and/or 1 yr post-TKA). It is not known if early gains in functional mobility will positively impact muscle cell function.
5. We expect to show that quality of life (as measured by instruments such as VR-12) will be significantly increased with EAA. It is not known to what extent the above positive gains will have on longer-term (6 mo and 1 yr) quality of life.

We expect each of the above to stimulate and be transformative. EAA supplements are inexpensive ($800/patient or $16/day), are well tolerated, and can be implemented immediately.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 50-80 years.
* Primary TKA surgery.

Exclusion Criteria:

1. Previous TKA and/or total hip arthroplasty surgery (older subjects).
2. Dementia or related mental issues that may potentially put the subject at risk as determined by the surgeon.
3. Untreated endocrine disease (Hypo/Hyperthyroidism, Addison's or Cushing's syndrome, etc.).
4. Significant heart, liver, kidney, blood, or respiratory disease.
5. Peripheral vascular disease.
6. Active cancer.
7. Recent (within 6 months) treatment with anabolic steroids.
8. Alcohol or drug abuse.
9. Inability to have MRI

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Oregon, Eugene, Oregon
  - Slocum Center for Orthopedics and Sports Medicine, Eugene, Oregon

REFERENCES:
- [Result] Dreyer HC, Owen EC, Strycker LA, Smolkowski K, Muyskens JB, Kirkpatrick TK, Christie AD, Kuehl KS, Lantz BA, Shah SN, Mohler CG, Jewett BA. Essential Amino Acid Supplementation Mitigates Muscle Atrophy After Total Knee Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial. JB JS Open Access. 2018 Jun 4;3(2):e0006. doi: 10.2106/JBJS.OA.18.00006. eCollection 2018 Jun 28. PMID 30280129
- [Result] Muyskens JB, Foote DM, Bigot NJ, Strycker LA, Smolkowski K, Kirkpatrick TK, Lantz BA, Shah SN, Mohler CG, Jewett BA, Owen EC, Dreyer HC. Cellular and morphological changes with EAA supplementation before and after total knee arthroplasty. J Appl Physiol (1985). 2019 Aug 1;127(2):531-545. doi: 10.1152/japplphysiol.00869.2018. Epub 2019 Jul 25. PMID 31343947
- [Result] Muyskens JB, Hocker AD, Turnbull DW, Shah SN, Lantz BA, Jewett BA, Dreyer HC. Transcriptional profiling and muscle cross-section analysis reveal signs of ischemia reperfusion injury following total knee arthroplasty with tourniquet. Physiol Rep. 2016 Jan;4(1):e12671. doi: 10.14814/phy2.12671. PMID 26733251
- [Result] Dreyer HC. Tourniquet Use During Knee Replacement Surgery May Contribute to Muscle Atrophy in Older Adults. Exerc Sport Sci Rev. 2016 Apr;44(2):61-70. doi: 10.1249/JES.0000000000000076. PMID 26829246
- See also: Muscle Physiology Lab at the University of Oregon — http://muscle.uoregon.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both aims will target older adults, ages 50 - 80 years for have elected to undergo primary total knee arthroplasty performed at PeaceHealth Sacred Heart Medical Center at RiverBend by Dr. Jewett, Lantz, Mohler or Shah. Between 2005-2010, they performed a total 2,066 TKAs. Of those, 1,406 of the patients were between 50-80 years of age (68%). A total of 120 subjects will be enrolled in the two study aims.
Groups:
- Essential Amino Acids (EAA): Aim 1: Twice-daily ingestion of 20 g of EAA for 1 wk before through 6 wk after TKA.
  Supplement composition for the EAAs: histidine, 2.2 g (11% of total); isoleucine, 2.0 g (10%); leucine, 3.6 g (18%); lysine, 3.2 g (16%); methionine, 0.6 g (3%); phenylalanine, 3.2 g (16%); threonine, 2.8 g (14%); and valine, 2.4 g (12%).
  Aim 2: Twice-daily ingestion of 23 g of EAA for 1 wk before through 6 wk after TKA.
  Supplement composition for the EAAs: histidine, 1.28 g (5% of total); isoleucine, 1.8 g (8%); leucine, 7.4 g (32%); lysine, 3.6 g (15%); methionine, 1.76 g (8%); phenylalanine, 3.1 g (13%); threonine, 1.9 g (8%); valine, 2.08 g (9%); and tryptophan, 0.5 g (2%).
  Essential Amino Acids (EAA): Twice daily ingestion of 20 or 23 grams of EAA for 7 days leading up to surgery and continuing for 6 weeks after surgery [surgery = primary total knee arthroplasty]
- Placebo (Alanine): Aim 1: Twice-daily ingestion of 20 g of Alanine (Non-essential amino acid) for 1 wk before through 6 wk after TKA.
  The placebo supplement consists of 20 g (100%) alanine.
  Aim 2: Twice-daily ingestion of 23 g of Alanine (Non-essential amino acid) for 1 wk before through 6 wk after TKA.
  The placebo supplement consists of 23 g (100%) alanine.
  Placebo (Alanine): Twice daily ingestion of 20 or 23 grams Placebo (alanine) for 7 days leading up to surgery and continuing for 6 weeks after surgery [surgery = primary total knee arthroplasty]
Period: Overall Study
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Started | 31 | 36
Completed | 19 | 20
Not Completed | 12 | 16

BASELINE CHARACTERISTICS:
Population: 31 subjects in EAA group began study and 19 completed study. 36 subjects in placebo group began study and 20 completed study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine) | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.95 (5.90) | 63.90 (5.37) | 64.41 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
MRI Quadriceps Involved Leg [Mean (Standard Deviation); unit: AU] — MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra to measure muscle volume in Arbitrary Units (AU). Low values = low volume. High values = higher volume.
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra (UO Lewis Center for Neuroimaging).
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  AU | 48.66 (14.62) | 44.81 (13.82) | 46.63 (14.14)
MRI Quadriceps Contralateral Leg [Mean (Standard Deviation); unit: AU] — MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra to measure muscle volume in Arbitrary Units (AU). Low values = low volume. High values = higher volume.
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra (UO Lewis Center for Neuroimaging).
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  AU | 55.49 (16.43) | 49.98 (13.64) | 52.59 (15.08)
MRI Hamstrings Involved Leg [Mean (Standard Deviation); unit: AU] — MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra to measure muscle volume in Arbitrary Units (AU). Low values = low volume. High values = higher volume.
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra (UO Lewis Center for Neuroimaging).
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  AU | 69.32 (17.65) | 63.86 (14.90) | 66.52 (16.32)
MRI Hamstrings Contralateral Leg [Mean (Standard Deviation); unit: AU] — MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra to measure muscle volume in Arbitrary Units (AU). Low values = low volume. High values = higher volume.
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra (UO Lewis Center for Neuroimaging).
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  AU | 69.37 (18.25) | 63.64 (14.88) | 66.43 (16.64)
Daily Physical Activity [Mean (Standard Deviation); unit: kcal/day] | 408.15 (192.47) | 319.71 (254.78) | 361.60 (228.82)
Handgrip Strength [Mean (Standard Deviation); unit: kg] | 29.95 (10.42) | 28.35 (8.44) | 28.64 (9.34)
Short Physical Performance Battery [Mean (Standard Deviation); unit: units on a scale] | 3.89 (0.32) | 4.00 (0.00) | 3.95 (0.22)
Timed Up and Go [Mean (Standard Deviation); unit: seconds] | 9.88 (2.02) | 11.40 (3.05) | 10.66 (2.68)
4-Meter Walk [Mean (Standard Deviation); unit: seconds] | 3.89 (0.32) | 3.80 (0.41) | 3.85 (0.37)
Stair Climb Up [Mean (Standard Deviation); unit: seconds] | 8.09 (2.40) | 9.45 (4.92) | 8.79 (3.91)
Stair Climb Down [Mean (Standard Deviation); unit: seconds] | 8.03 (2.92) | 10.70 (4.74) | 9.40 (4.13)
6-Minute Walk [Mean (Standard Deviation); unit: meters] | 511.10 (77.29) | 488.30 (101.96) | 499.41 (90.34)
KOOS Symptoms [Mean (Standard Deviation); unit: units on a scale] | 54.13 (18.98) | 50.00 (16.31) | 52.01 (17.55)
KOOS Pain [Mean (Standard Deviation); unit: units on a scale] | 51.18 (15.73) | 53.06 (14.56) | 52.14 (14.97)
KOOS Function Daily Living [Mean (Standard Deviation); unit: units on a scale] | 66.01 (15.00) | 60.67 (15.60) | 63.34 (15.34)
KOOS Function Sports/Recreation [Mean (Standard Deviation); unit: units on a scale] | 27.90 (20.43) | 30.00 (26.36) | 28.97 (23.37)
KOOS Knee-Related Quality of Life [Mean (Standard Deviation); unit: units on a scale] | 30.26 (13.70) | 24.01 (17.46) | 27.14 (15.80)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] | 3.42 (4.57) | 4.10 (3.78) | 3.77 (4.15)
PCS12 [Mean (Standard Deviation); unit: units on a scale] | 33.17 (9.55) | 33.41 (9.08) | 33.30 (9.15)
MCS12 [Mean (Standard Deviation); unit: units on a scale] | 55.48 (10.60) | 57.23 (7.26) | 56.43 (8.85)

OUTCOME MEASURES:

1. Primary Outcome: MRI Quadriceps Involved Leg
Description: MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra to measure muscle volume in Arbitrary Units (AU). Low values = low volume. High values = higher volume.
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
  MRI of the bilateral lower extremities was performed utilizing a Siemens 3T Skyra (UO Lewis Center for Neuroimaging).
  Dixon pulse sequence optimized for imaging near metal implants was used to capture T1-weighted, water, and fat images of the mid-thigh region.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
AU | 43.87 (12.08) | 38.31 (10.69)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .03, ANCOVA

2. Primary Outcome: MRI Quadriceps Contralateral Leg
Description: as for outcome 1
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
AU | 54.41 (15.50) | 46.44 (13.16)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .01, ANCOVA

3. Primary Outcome: MRI Hamstrings Involved Leg
Description: as for outcome 1
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
AU | 63.76 (14.88) | 55.93 (13.01)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .04, ANCOVA

4. Primary Outcome: MRI Hamstrings Contralateral Leg
Description: as for outcome 1
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
AU | 67.50 (16.33) | 58.75 (13.65)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .01, ANCOVA

5. Secondary Outcome: Daily Physical Activity
Description: Average daily calories expended in physical activity calculated from accelerometer data
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
kcal/day | 265.67 (151.43) | 196.54 (80.34)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .12, ANCOVA

6. Secondary Outcome: Handgrip Strength
Description: Maximum isometric strength of the hand and forearm muscles measured by a handgrip dynamometer
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
kg | 30.74 (10.61) | 28.03 (8.37)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .03, ANCOVA

7. Secondary Outcome: Short Physical Performance Battery
Description: Short Physical Performance Battery. Minimum = 0. Maximum = 11. 0 representing extreme problems and 11 is no problems. The higher the score the better the outcome.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
units on a scale | 3.95 (0.23) | 3.90 (0.31)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .71, ANCOVA

8. Secondary Outcome: Timed Up and Go
Description: Time from a seated position to walk forward 3 meters, turn around, walk back 3 meters, and sit down again
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
seconds | 9.87 (1.92) | 10.90 (3.71)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .76, ANCOVA

9. Secondary Outcome: 4-Meter Walk
Description: Time from a standing position to walk 4 meters through the finish line
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
seconds | 3.89 (0.32) | 3.90 (0.31)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .40, ANCOVA

10. Secondary Outcome: Stair Climb Up
Description: Time to climb up 11 steps
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
seconds | 7.95 (2.80) | 8.64 (3.40)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .97, ANCOVA

11. Secondary Outcome: Stair Climb Down
Description: Time to climb down 11 steps
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
seconds | 8.12 (3.22) | 9.53 (4.57)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .89, ANCOVA

12. Secondary Outcome: 6-Minute Walk
Description: Total distance walked in 6 minutes
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
meters | 464.56 (139.40) | 477.02 (103.96)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .48, ANCOVA

13. Secondary Outcome: KOOS Symptoms
Description: Knee Injury and Osteoarthritis Outcome Score measuring patients' overall opinions about knee and associated problems.
  Minimum = 0. Maximum = 100. 0 representing extreme problems and 100 representing no problems.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
scores on a scale | 68.80 (12.36) | 56.99 (15.70)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .02, ANCOVA

14. Secondary Outcome: KOOS Pain
Description: Knee Injury and Osteoarthritis Outcome Score measuring patients' opinions about knee-specific pain; 0-100 Minimum = 0. Maximum = 100. 0 representing extreme problems and 100 representing no problems.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
scores on a scale | 68.71 (8.97) | 64.77 (14.87)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .29, ANCOVA

15. Secondary Outcome: KOOS Function Daily Living
Description: Knee Injury and Osteoarthritis Outcome Score measuring patients' opinions about knee-specific function in daily life; 0-100 Minimum = 0. Maximum = 100. 0 representing extreme problems and 100 representing no problems.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
score on a scale | 81.41 (10.52) | 76.16 (12.10)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .33, ANCOVA

16. Secondary Outcome: KOOS Function Sports/Recreation
Description: Knee Injury and Osteoarthritis Outcome Score measuring patients' opinions about knee-specific function in sport and recreation; 0-100 Minimum = 0. Maximum = 100. 0 representing extreme problems and 100 representing no problems.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
score on a scale | 44.21 (27.70) | 37.90 (22.87)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .30, ANCOVA

17. Secondary Outcome: KOOS Knee-Related Quality of Life
Description: Knee Injury and Osteoarthritis Outcome Score measuring patients' opinions about knee-related quality of life; 0-100 Minimum = 0. Maximum = 100. 0 representing extreme problems and 100 representing no problems.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
score on a scale | 51.74 (17.78) | 50.33 (16.33)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .98, ANCOVA

18. Secondary Outcome: PHQ-9
Description: Patient Health Questionnaire depression module measuring depression symptom severity; 0-27.
  0 is minimum and 27 is maximum. Lower score is less depression symptoms. Higher score is high depression symptoms.
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
score on a scale | 4.68 (3.70) | 3.68 (2.75)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .18, ANCOVA

19. Secondary Outcome: PCS12
Description: Veterans Rand 12-item Health Survey Physical Component Summary norm-referenced score reflecting physical health-related quality of life.
  Minimum = 0. Maximum = 100. 0 representing extreme problems and 100
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
score on a scale | 37.55 (8.83) | 35.48 (7.27)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .52, ANCOVA

20. Secondary Outcome: MCS12
Description: Veterans Rand 12-item Health Survey Mental Component Summary norm-referenced score reflecting mental health-related quality of life.
  Minimum = 0. Maximum = 100. 0 representing extreme problems and 100
Time Frame: 6 weeks after baseline
Population: enrolled participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
Number analyzed (Participants) | 19 | 20
score on a scale | 52.11 (11.01) | 54.76 (11.60)
Statistical Analysis 1: Comparison: Essential Amino Acids (EAA) vs Placebo (Alanine); Test type: Other; p = .81, ANCOVA

ADVERSE EVENTS:
Time Frame: baseline to 6 weeks
Description: The study assessed the effectiveness of FDA-approved over-the-counter supplements, which did not cause any participants to be at risk for Serious Adverse Events, All-Cause Mortality, and Other Adverse Events.
Arm/Group | Essential Amino Acids (EAA) | Placebo (Alanine)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/31 | 4/36
Other Adverse Events (participants affected / at risk) | 0/31 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essential Amino Acids (EAA) (N=31) | Placebo (Alanine) (N=36)
Nausea (General disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT02145949/Prot_SAP_ICF_000.pdf